CLINICAL TRIAL: NCT06305455
Title: Change in the Resistance Profile of Escherichia Coli in Infections of Community Origin: The Importance of Antimicrobial Stewardship
Brief Title: Resistance Profile of Escherichia Coli in Infections of Community Origin: The Importance of Antimicrobial Stewardship
Status: Not yet recruiting | Type: Observational
Sponsor: José Raimundo Araujo de Azevedo (Other)
Responsible Party: Sponsor-Investigator, José Raimundo Araujo de Azevedo, Clinical Researcher, Hospital Sao Domingos
Organization: Hospital Sao Domingos (Other)
Other Study IDs: HSD135
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Antimicrobial Resistance
Keywords: antimicrobial resistance; Escherichia coli ESBL; antimicrobial stewardship; community infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Escherichia coli ESBL — To evaluate the change in the resistance profile of infections of community origin caused by Escherichia coli, isolated from any culture material in patients admitted to the intensive care unit of a tertiary hospital.

SUMMARY:
The main objective of the study is to describe the antimicrobial resistance profile of E. coli isolated in patients from the community - defined as those with cultures collected within 48 hours of hospital admission - and admitted to the intensive care unit.

DETAILED DESCRIPTION:
Background: The growing antimicrobial resistance in bacterial pathogens represents a severe public health problem. Isolation of Escherichia coli ESBL has been identified more frequently over the years due to the worldwide dissemination of strains with this phenotypic profile. The ICU has a fully functioning Antimicrobial Stewardship team, with data managed daily. Thus, the investigators identified increasing E. coli ESBL isolates resistant to standard empiric antimicrobial therapy in community-based severe infections.

Purpose: The choice of empirical antimicrobial therapy is an increasingly present challenge in clinical practice, often determining the outcome of critically ill patients. As this is a highly relevant topic in managing this patient profile, antimicrobial stewardship protocols are essential in health services, enabling continuous community monitoring of emerging resistance profiles. The justification for this study is based on the possibility of adding knowledge on the topic, aiming to add to the global theoretical collection and alert about the locoregional occurrence of changes in the bacterial resistance profile.

Objectives: The main objective of the study is to describe the antimicrobial resistance profile of E. coli isolated in patients from the community - defined as those with cultures collected within 48 hours of hospital admission - and admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* All 18 years and old patients admitted to the ICU
* Positive cultures for E. coli
* Any sample collected within 48 hours of hospital admission

Exclusion Criteria:

* Lack of necessary data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe Escherichia coli infections, isolated from any culture material collected within less than 48 hours of hospital admission, admitted to the intensive care unit of a tertiary hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Escherichia coli resistance | 24 months
  The main objective of the study is to describe the antimicrobial resistance profile of E. coli isolated in patients from the community admitted to the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: RODRIGO AZEVEDO, MD, PhD, Study Director — Hospital São Domingos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenreich W, Rudel T, Heesemann J, Goebel W. Link Between Antibiotic Persistence and Antibiotic Resistance in Bacterial Pathogens. Front Cell Infect Microbiol. 2022 Jul 19;12:900848. doi: 10.3389/fcimb.2022.900848. eCollection 2022. PMID 35928205
- [Result] Zhu DM, Li QH, Shen Y, Zhang Q. Risk factors for quinolone-resistant Escherichia coli infection: a systematic review and meta-analysis. Antimicrob Resist Infect Control. 2020 Jan 9;9(1):11. doi: 10.1186/s13756-019-0675-3. eCollection 2020. PMID 31938541
- [Result] Castanheira M, Deshpande LM, Mendes RE, Canton R, Sader HS, Jones RN. Variations in the Occurrence of Resistance Phenotypes and Carbapenemase Genes Among Enterobacteriaceae Isolates in 20 Years of the SENTRY Antimicrobial Surveillance Program. Open Forum Infect Dis. 2019 Mar 15;6(Suppl 1):S23-S33. doi: 10.1093/ofid/ofy347. eCollection 2019 Mar. PMID 30895212
- [Result] Canton R, Gijon D, Ruiz-Garbajosa P. Antimicrobial resistance in ICUs: an update in the light of the COVID-19 pandemic. Curr Opin Crit Care. 2020 Oct;26(5):433-441. doi: 10.1097/MCC.0000000000000755. PMID 32739970
- [Result] Kim JY, Yum Y, Joo HJ, An H, Yoon YK, Kim JH, Sohn JW. Impact of antibiotic usage on extended-spectrum beta-lactamase producing Escherichia coli prevalence. Sci Rep. 2021 Jun 22;11(1):13024. doi: 10.1038/s41598-021-91332-x. PMID 34158540